CLINICAL TRIAL: NCT04819269
Title: Tivanisiran for Dry Eye in Subjects With Sjögren's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYL1001_V
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Disease; Sjögren Syndrome
Keywords: oligonucleotide; siRNA; keratoconjunctivitis sicca; SYL1001
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tivanisiran sodium ophthalmic solution (Active Comparator)
  Interventions: Drug: Tivanisiran sodium ophthalmic solution
- Vehicle ophthalmic solution (Placebo Comparator)
  Interventions: Drug: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: Tivanisiran sodium ophthalmic solution — 1 drop in the affected eye(s) once daily
  Arms: Tivanisiran sodium ophthalmic solution
Drug: Vehicle ophthalmic solution — 1 drop in the affected eye(s) once daily
  Arms: Vehicle ophthalmic solution

SUMMARY:
This study will examine the efficacy and safety of tivanisiran sodium eye drops versus vehicle after a 2-week run-in phase when dosed once daily for 3 months in subjects with signs and symptoms of dry eye disease (DED) due to Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or a female aged ≥ 18 years
* Have given their written consent to participate in the study
* Use of artificial tears (AT), autologous serum or specific dry eye medications during the last 6 months prior to the selection
* Willing to not use AT or autologous serum for the study duration
* VAS scale for Dry Eye Symptom Score ≥ 40
* Total CFS ≥ 5
* Schirmer's test with anesthesia < 10 mm/5min
* Patients with Sjögren Syndrome

Exclusion Criteria:

* Any concomitant treatment or prior ocular procedure or surgery, or alteration of the dose of systemic medications at the time of entry into the study
* Use of contact lenses during the study
* Significant Eye diseases according to investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Corneal Fluorescein Staining (CFS) scale [0-3]. Higher scores mean disease worsening. | 85 days
Change from baseline in Dry Eye Symptom scale [0-100]. Higher scores mean disease worsening. | 85 days

CONTACTS AND LOCATIONS:
Locations (44):
- United States (38):
  - Sylentis Investigative Site, Birmingham, Alabama
  - Sylentis Investigative Site, Dothan, Alabama
  - Sylentis Investigative Site, Scottsdale, Arizona
  - Sylentis Investigative Site, Garden Grove, California
  - Sylentis Investigative Site, Glendale, California
  - Sylentis Investigative Site, Los Angeles, California
  - Sylentis Investigative Site, Newport Beach, California
  - Sylentis Investigative Site, Rancho Cordova, California
  - Sylentis Investigative Site, San Diego, California
  - Sylentis Investigative Site, Torrance, California
  - Sylentis Investigative Site, Aurora, Colorado
  - Sylentis Investigative Site, Colorado Springs, Colorado
  - Sylentis Investigative Site, Littleton, Colorado
  - Sylentis Investigative Site, Jacksonville, Florida
  - Sylentis Investigative Site, Largo, Florida
  - Sylentis Investigative Site, Miami, Florida
  - Sylentis Investigative Site, Ormond Beach, Florida
  - Sylentis Investigative Site, Tampa, Florida
  - Sylentis Investigative Site, Atlanta, Georgia
  - Sylentis Investigative Site, Morrow, Georgia
  - Sylentis Investigative Site, Carmel, Indiana
  - Sylentis Investigative Site, Waltham, Massachusetts
  - Sylentis Investigative Site, Ypsilanti, Michigan
  - Sylentis Investigative Site, Kansas City, Missouri
  - Sylentis Investigative Site, St Louis, Missouri
  - Sylentis Investigative Site, Washington, Missouri
  - Sylentis Investigative Site, Asheville, North Carolina
  - Sylentis Investigative Site, High Point, North Carolina
  - Sylentis Investigative Site, Fargo, North Dakota
  - Sylentis Investigative Site, Cleveland, Ohio
  - Sylentis Investigative Site, Columbus, Ohio
  - Sylentis Investigative Site, Cranberry Township, Pennsylvania
  - Sylentis Investigative Site, Rapid City, South Dakota
  - Sylentis Investigative Site, Memphis, Tennessee
  - Sylentis Investigative Site, Nashville, Tennessee
  - Sylentis Investigative Site, El Paso, Texas
  - Sylentis Investigative Site, Houston, Texas
  - Sylentis Investigative Site, Falls Church, Virginia
- Spain (6):
  - Sylentis Investigative Site, Pamplona, Navarre
  - Sylentis Investigative Site, Barcelona
  - Sylentis Investigative Site, Madrid
  - Sylentis Investigative Site, Seville
  - Sylentis Investigative Sites, Valladolid
  - Sylentis Investigative Site, Zaragoza